CLINICAL TRIAL: NCT03793582
Title: Impact of Obstructive Sleep Apnea on Outcomes in Acute Coronary Syndrome
Brief Title: Impact of OSA on Outcomes in Acute Coronary Syndrome
Acronym: ISAACS
Status: Completed | Type: Observational
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Dennis Auckley, MD, Professor of Medicine, MetroHealth Medical Center
Other Study IDs: IRB16-00812
Record Dates: First submitted 2018-11-21; First posted 2019-01-04 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: OSA; ACS - Acute Coronary Syndrome; Major Adverse Cardiac Events
Keywords: OSA; ACS (Acute Coronary Syndrome); MACE (Major Adverse Cardiac Events)
MeSH Terms: conditions — Acute Coronary Syndrome; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Study group: All subjects agreeing to participate and meeting inclusion criteria but not meeting exclusion criteria
  Interventions: Diagnostic Test: ApneaLink Type III portable sleep study

INTERVENTIONS:
Diagnostic Test: ApneaLink Type III portable sleep study — Type III portable sleep study

SUMMARY:
Elucidating the effects of obstructive sleep apnea (OSA) on cardiovascular outcomes in acute coronary syndrome (ACS) is crucial in risk assessments and therapeutic recommendations for affected individuals. Although large epidemiological studies have reported an association between OSA and both coronary heart disease (CHD) and heart failure (HF), its effect on outcomes in ACS is still unclear. In contrast to previous theories attributing causation to OSA, recent studies have hypothesized a cardio protective role of OSA. Repetitive hypoxemic episodes noted in OSA may lead to myocardial ischemic preconditioning, possibly by increasing coronary collateral vessel recruitment, conferring protection from acute coronary events. We propose a prospective, observational, single center study in patients presenting with ACS, including ST segment elevation (STEMI), non-ST segment elevation (NSTEMI) and unstable angina who undergo coronary revascularization to determine the impact of OSA on clinical outcomes after ACS. Adult patients above age 18 years who present with myocardial infarction are eligible. Recruited patients will undergo an overnight sleep study using a level III portable diagnostic device before hospital discharge. The sleep tracings will be analyzed and audited by a certified sleep physician. The patients will be divided into 2 groups based on apnea-hypopnea index (AHI): OSA (AHI ≥ 15) and non-OSA (AHI < 15) groups. The primary end points of this study were in-hospital, 30 day and 6 month major adverse cardiovascular events (MACE), defined as a composite endpoint of cardiovascular death, non-fatal MI, stroke and the need for unplanned repeat revascularization. Secondary endpoints include individual MACE outcomes of cardiovascular death, non-fatal MI, stroke, need for unplanned repeat revascularization, heart failure requiring hospitalization, and all-cause mortality.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is very common in middle aged adults. Using a polysomnography (PSG) derived definition, defined as an apnea hypopnea index (AHI) of >5, it occurs in 20-30 % of males and 10-15 % of females in North America. Various large epidemiological studies have established a close relationship between OSA and cardiovascular disease including coronary heart disease (CHD), heart failure, atrial fibrillation, and stroke. Potential mechanisms including endothelial dysfunction/ systemic inflammation, sympathetic activation, metabolic dysregulation, and mechanical load effects during respiratory events have been implicated for this relationship. However, in contrast to previous literature, more recent studies have also explored a cardio protective role of OSA. Repetitive hypoxemic episodes noted in OSA may lead to myocardial ischemic preconditioning, conferring protection in the form of a smaller myocardial infarct size, lower rates of cardiac arrhythmias, heart failure, and thereby, cardiovascular mortality. Animals exposed to intermittent hypoxia prior to ischemic insult experience significantly reduced infarct sizes when compared to animals not exposed to intermittent hypoxemia. Whether a similar effect exists in humans is still unclear. Recent research indicates better coronary collateral flow in OSA compared to control subjects presenting with acute coronary syndrome (ACS), which potentially could explain a cardioprotective role. Others have reported variable outcomes of coronary plaque burden and lesion complexity, restenosis and target vessel revascularization, serological markers such as troponin T, high sensitivity-C reactive protein (hs-CRP) and N-terminal pro brain natriuretic peptide (NT-proBNP), and major adverse cardiovascular events (MACE) in OSA vs. control subjects. Further, some of these early reports were limited by available devices, technology and methodology of the era. The objective of this study is to examine the prognostic role of OSA in patients with acute coronary syndrome (ACS). We tested the hypothesis whether OSA predicts subsequent MACE in patients undergoing percutaneous coronary intervention.

Methods This is a prospective, single center, observational study of patients presenting with ACS, including ST segment elevation (STEMI), non-ST segment elevation (NSTEMI) and unstable angina who undergo coronary revascularization at our tertiary care center. A total of 160 adult patients above age 18 years who meet our inclusion/ exclusion criteria will be enrolled. The estimated duration for this study is 2017-2018.

Prospective eligible patients who present for treatment for ACS at our institution in the study period will be approached for recruitment. Exclusion criteria for the study include: pregnancy, post-cardiac arrest patients, diagnosis of medical conditions associated with predicted survival of < 6 months, need for tracheostomy and prolonged mechanical ventilation, prior treatment for sleep disordered breathing and unavailable sleep data (due to death, no informed consent, uncooperative subject, technical difficulties, miscellaneous).

All subjects or their legally authorized representatives must provide written informed consent before any study-related procedure can be conducted. All recruited patients will undergo a level III sleep study within 48 to 72 hours prior to discharge. The patients will then be separated into OSA (AHI≥15 events/ h) and non-OSA (AHI<15) groups based on AHI.

There will be no financial incentive offered to patients. All recruited patients will be treated according to Declaration of Helsinki and amendments, World Medical Association Declaration of Helsinki - Ethical Principles for Medical Research Involving Human Subjects and standard clinical guidelines.

Study data will be collected and managed using REDCap electronic data capture tools hosted at MetroHealth Medical Center. REDCap (Research Electronic Data Capture) is a secure, web-based application designed to support data capture for research studies, providing: 1) an intuitive interface for validated data entry; 2) audit trails for tracking data manipulation and export procedures; 3) automated export procedures for seamless data downloads to common statistical packages; and 4) procedures for importing data from external sources.

Study Endpoints Baseline patient information will be collected prospectively at presentation for the index hospitalization for acute MI including: demographic information, cardiovascular risk factors, medical conditions, current medications, and relevant laboratory test values. The primary end point of this study were in-hospital, 30 day major adverse cardiac events (MACE), defined as a composite endpoint of cardiovascular death, non-fatal MI, stroke and the need for unplanned repeat revascularization. Secondary endpoints include 6 month major adverse cardiac events (MACE), individual MACE cardiovascular death, non-fatal MI, stroke, need for unplanned repeat revascularization, ST segment resolution (STR), heart failure requiring hospitalization, and all-cause mortality.

Percutaneous Coronary Intervention Primary PCI will be performed according to the standard clinical practice. There are no restrictions to the usage of pharmacologic and device strategies during PCI. PCI is defined as any intervention to a major epicardial coronary artery with a significant stenosis based on ≥70%-diameter narrowing on visual estimation (≥50% for left main) and/or fulfilling physiological criteria for revascularization (i.e., fractional flow reserve ≤0.80, intravascular ultrasound-IVUS). Angiographic findings including TIMI flow and ST resolution will be obtained as standard of care by the cardiology team.

Echocardiography Comprehensive Transthoracic 2D and Doppler echocardiography using commercially available echocardiography machines will be obtained during hospitalization. Standard parasternal, apical, and subcostal views will be obtained with the subject in a left lateral recumbent position. Images were stored digitally and on VHS videotape, which were subsequently analyzed. All measurements will be made according to American Society of Echocardiography Guidelines.

Overnight Sleep Study All sleep studies will be conducted using a Resmed ApneaLink Air standardized level III portable diagnostic device (ResMed Corporation, Poway, California). Although limited by its inability to identify sleep stages and lack of an objective measurement of sleep duration, this device has been validated for use against in-laboratory polysomnography with sensitivity and specificity around 91% and 95% at an AHI value of ≥15/ hour, respectively. Outputs recorded from the portable diagnostic device include nasal airflow (nasal pressure transducer), thoraco-abdominal movements (inductive respiratory band), arterial oxygen saturation (pulse oximetry), and snoring episodes (derived from the integrated pressure transducer). All studies will be manually scored and analyzed by a certified sleep physician. To ensure the accuracy and consistency of scorings, a second sleep physician will audit the studies.

The primary measure of the sleep study will be the AHI, quantified as the total number of apneas and hypopneas per hour of sleep. The respiratory event scoring will be performed according to the American Academy of Sleep Medicine guidelines.

Standardized Obstructive Sleep Apnea Questionnaire Administration During hospitalization for acute MI, recruited patients will be administered the STOP-BANG Questionnaire, Berlin Questionnaire (BQ) and Epworth Sleepiness Scale (ESS) by face-to-face interviews by an investigator.

Referral to Sleep Clinic All patients diagnosed with OSA during this study will be referred to the Sleep Clinic at MetroHealth Medical Center for further evaluation and treatment. Relevant sleep study data will be made available to patients and clinicians.

Follow up Patient data will be collected at 30-days and 6 months to record outcomes.

Sample- Size Calculation According to previous study, 23.5% of patients with OSA, based on an AHI ≥10 are expected to have adverse MACE after undergoing PCI for ACS, whereas only 5.3% non-OSA patients experienced these events. Based on 85% power and a significance level of 5%, the required sample size is 130 (OSA, n=65; non-OSA, n=65). Given that an estimated 20% of the sleep studies may not be successful (due to premature device removal by the patients or technical errors), a minimum of 162 recruited patients is needed. The projected sample size of 160 participants will provide sufficient power to test the primary hypothesis.

ELIGIBILITY:
Inclusion Criteria:

Patients presenting with:

* Acute coronary syndrome, including:

  * ST segment elevation (STEMI)
  * non-ST segment elevation (NSTEMI)
  * unstable angina
* Who undergo coronary revascularization at our tertiary care center .

Exclusion Criteria:

* Pregnancy
* Post-cardiac arrest patients
* Diagnosis of medical conditions associated with predicted survival of < 6 months
* Need for tracheostomy and prolonged mechanical ventilation
* Prior treatment for sleep disordered breathing and unavailable sleep data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients admitted to MetroHealth Medical Center with acute coronary syndrome (ACS) that meet inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
MACE | 30 days
  Number of patients with major adverse cardiac events (MACE)

SECONDARY OUTCOMES:
Individual MACE outcomes | 30 days and 6 months
  Number of patients with nonfatal MI, CVA, unplanned revascularization, CHF, CV death, all-cause death
MACE | 6 months
  Number of patients with major adverse cardiac events

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Auckley, MD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] Shahar E, Whitney CW, Redline S, Lee ET, Newman AB, Nieto FJ, O'Connor GT, Boland LL, Schwartz JE, Samet JM. Sleep-disordered breathing and cardiovascular disease: cross-sectional results of the Sleep Heart Health Study. Am J Respir Crit Care Med. 2001 Jan;163(1):19-25. doi: 10.1164/ajrccm.163.1.2001008. PMID 11208620
- [Background] Hla KM, Young T, Hagen EW, Stein JH, Finn LA, Nieto FJ, Peppard PE. Coronary heart disease incidence in sleep disordered breathing: the Wisconsin Sleep Cohort Study. Sleep. 2015 May 1;38(5):677-84. doi: 10.5665/sleep.4654. PMID 25515104
- [Background] Yumino D, Tsurumi Y, Takagi A, Suzuki K, Kasanuki H. Impact of obstructive sleep apnea on clinical and angiographic outcomes following percutaneous coronary intervention in patients with acute coronary syndrome. Am J Cardiol. 2007 Jan 1;99(1):26-30. doi: 10.1016/j.amjcard.2006.07.055. Epub 2006 Nov 2. PMID 17196456
- [Background] Hein T, Loo G, Ng WY, Tai BC, Kajiya T, Tan A, Khoo SM, Chan M, Low AF, Chia BL, Richards M, Lee CH. Relationship between apnoea-hypopnoea index and angiographic coronary disease phenotypes in patients presenting with acute myocardial infarction. Acute Card Care. 2013 Jun;15(2):26-33. doi: 10.3109/17482941.2012.741249. PMID 23738622